CLINICAL TRIAL: NCT04005482
Title: Blood Pressure During Rate Control in Patients With Tachycardic Atrial Fibrillation at the Emergency Department
Acronym: BPIRCTPTAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Hans Domanovits, Principal Investigator, Medical University of Vienna
Other Study IDs: MUVienna 1568/2014
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Heart Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rate control — Rate control according to the Atrial fibrillation - ESC Guidelines 2016

SUMMARY:
The aim of this study is to analyse blood pressure during rate control therapy in patients with tachycardic atrial fibrillation in a real-world emergency cohort.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the primary clinical problem in 3.3% to 10.0 % emergency department (ED) admissions. Rate control is an integral part of the management of symptomatic tachycardic AF patients.

According to the recent guidelines beta-blockers, digoxin, the calcium channel blockers diltiazem and verapamil, amiodarone or combination therapy should be considered for rate control. Haemodynamic side-effects in particular hypotension may occur. Heart rate and blood pressure behavior in an ED population during rate control therapy in patients with tachycardic atrial fibrillation will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Atrial fibrillation or atrial flutter and heart rate ≥ 110 bpm
* Indication for rate control
* Informed consent

Exclusion Criteria:

• Inclusion criteria not met

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include all patients admitted to the Emergency Department of the Medical University Vienna with tachycardic AF receiving rate control therapy.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
Mean and maximum blood pressure difference between before (baseline) and during/after medication. | 20th July 2019 to 20th July 2021

CONTACTS AND LOCATIONS:
Overall Officials: Hans Domanovits, Prof., Study Director — Emergency Department, Medical University Vienna

IPD SHARING:
Plan to Share IPD: Undecided